CLINICAL TRIAL: NCT01188070
Title: Caregiver Stress: Interventions to Promote Health and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, ECorwin, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00032005; P01NR011587 (NIH)
Record Dates: First submitted 2010-06-14; First posted 2010-08-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Health Promotion
Keywords: Behavioral/Social; Cardiology; Clinical Laboratory Methods; Congestive Heart Failure; Heart Disease; Knowledge Dissemination; Lipids; Nursing; Health Promotion; Alzheimer's Disease/Dementia
MeSH Terms: conditions — Behavior; Heart Failure; Heart Diseases; Alzheimer Disease; Dementia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care Attention Control (Sham Comparator): Provision of printed educational material and attendance at one group session. This session will focus on nutrition education and flexibility and stretching.
  Interventions: Behavioral: Usual Care
- Psychoeducation plus exercise (Experimental): Psychoeducation intervention plus an individualized exercise program which will include monitored, individually-prescribed aerobic and resistance exercise.
  Interventions: Behavioral: Psycho-education plus physical exercise
- Psychoeducation (Active Comparator): Psychoeducational program to involve group sessions over consecutive weeks. The sessions will use the principles of adult learning, emphasizing active learning, group exercises and discussion, and coaching as well as brief talks to provide content. The curriculum will focus on the strengthening of caregiver self-efficacy through enhancement of knowledge and understanding, the acquisition, strengthening, and practice of caregiving skills, and the development of a more clinical or strategic outlook on the caregiving role.
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Usual Care — Educational materials
  Arms: Usual Care Attention Control
Behavioral: Psycho-education — Educational group sessions
  Arms: Psychoeducation
Behavioral: Psycho-education plus physical exercise — Psychoeducation intervention plus an individualized exercise program
  Arms: Psychoeducation plus exercise

SUMMARY:
More and more family members are providing care to their loved ones with prolonged and progressive illnesses. Chronic intense caregiving represents a situation of chronic stress, which takes a toll on one's mental and physical health including an increased risk for the development or worsening of heart disease. Identification of effective self-care interventions for family caregivers is warranted to improve their emotional wellbeing and minimize the harmful effects of chronic stress on the heart. This Program Project Grant aims to promote health and reduce cardiovascular risk in family caregivers (FCG) of persons with chronic illness. In two studies the investigators will test two interventions, psycho-education(ED) and physical exercise(EX), individually and in combination. The first study will target FCG of African American dementia patients; the second will focus on FCG of heart failure patients. Parallel designs, interventions and measures will create synergy as will integration of all data management and analyses within a Bio-behavioral Science and Measures Core. This Core will also provide high level guidance and interpretation of model testing resulting from analysis of the common data set. The combined de-identified data set will allow for elucidating the biological mechanisms of stress-induced cardiovascular risk, further developing the model, and stimulating future research, while the shared core support will provide substantial efficiency; neither could be achieved outside of a Program Project approach. These collective efforts will generate important data whereby future care can significantly enhance the lives of FCG and minimize their risk of cardiovascular disease, the number one cause of disability and death in the United States.

We hypothesize that FCGs who receive the combined PSYCHED+EX intervention will have better psychological functioning (lower levels of depressive symptoms, anxiety, and caregiver burden and higher levels of flourishing), behavioral outcomes (improved sleep quality and greater physical function), cardiovascular risk measures (improved resting heart rate, blood pressure, heart rate recovery, oxygen consumption, lipids, glucose, and inflammatory markers), neuroendocrine function (salivary cortisol) and overall health outcomes (improved function, muscle strength, and endurance) compared to psycho-education and usual care-attention control from baseline to six months later mediated by improvements in process outcomes (lower perceived stress and higher self-efficacy).

ELIGIBILITY:
Inclusion Criteria:

* Family caregiver defined as a spouse, partner or other adult family member living in the same house or in contact with a HF patient or dementia patient in a caregiver relationship at least 4 times/week for at least one hour or more.
* willing to participate
* English fluency
* ambulatory and physically able to engage in a structured low impact walking and upper body strength training program.
* self identify as African American for the Alzheimer FCG study

Exclusion Criteria:

* non sedentary (defined as engaging in > 30 minutes of moderately strenuous exercise 3 times or more a week)
* medical or physical condition that would preclude participation in the exercise component of the study (e.g., severe arthritis or mobility problems, uncontrolled hypertension or diabetes, renal insufficiency, or a history of angina with activity)
* current psychiatric comorbidity (alcohol or drug abuse/dependence, bipolar or psychotic disorder, suicidal ideation detected on the MINI screening tool)
* current smoker
* cognitive problems (BLESSED screen)
* ischemic changes or inappropriate BP changes on BL exercise (modified Balke) treadmill test
* on corticosteroids
* experiencing an acute inflammation at time of baseline or follow-up testing (this will result in rescheduling of testing if no other exclusion criteria apply)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Emotional outcomes | Baseline and 6 months
  Depression, Anxiety, Caregiver Burden, Flourishing
Behavioral Outcomes | Baseline and 6 months
  Physical Activity, Sleep Quality
Health Status | Baseline and 6 months
  Function, Muscle strength, endurance
Neuroendocrine | Frame Baseline and 6 months
  Salivary Cortisol
Cardiovascular Risk Outcomes | Baseline and 6 months
  Biochemical Markers (Inflammation Coagulation Insulin Resistance) Cardiovascular Reactivity & Risk

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Miller, MD, Principal Investigator — Emory University; Kenneth Hepburn, PhD, Study Chair — Emory University; Sandra Dunbar, DSN, Study Chair — Emory University; Monica Parker, MD, Study Chair — Emory University; Elizabeth J Corwin, PhD, Principal Investigator — Emory University School of Nursing
Locations (1):
- Emory Universtiy, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Corrigendum. J Appl Gerontol. 2020 Feb;39(2):NP1. doi: 10.1177/0733464818775576. Epub 2018 Apr 30. PMID 29708007
- [Derived] Gary R, Dunbar SB, Higgins M, Butts B, Corwin E, Hepburn K, Butler J, Miller AH. An Intervention to Improve Physical Function and Caregiver Perceptions in Family Caregivers of Persons With Heart Failure. J Appl Gerontol. 2020 Feb;39(2):181-191. doi: 10.1177/0733464817746757. Epub 2018 Jan 18. PMID 29347863